CLINICAL TRIAL: NCT01528709
Title: Aggressive Cholesterol Therapy to Inhibit Vein Graft Events (ACTIVE Trial): Does High-Dose Postoperative Statin Therapy Improve Graft Patency After Coronary Bypass?
Brief Title: Aggressive Cholesterol Therapy to Inhibit Vein Graft Events After CABG (ACTIVE Trial)
Acronym: ACTIVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boca Raton Regional Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Alexander Kulik, Cardiovascular Surgeon, Boca Raton Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011.02
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Results first posted 2018-08-09 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Saphenous Vein Graft Disease
Keywords: Statin,; CABG,; saphenous vein graft,; graft occlusion,; lipids
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-dose statin therapy (Experimental): Atorvastatin 80 mg daily
  Interventions: Drug: Atorvastatin 80 mg daily
- Moderate-dose statin therapy (Active Comparator): Atorvastatin 10 mg daily
  Interventions: Drug: Atorvastatin 10 mg daily

INTERVENTIONS:
Drug: Atorvastatin 80 mg daily — Atorvastatin 80 mg daily for 1 year
  Arms: High-dose statin therapy
Drug: Atorvastatin 10 mg daily — Atorvastatin 10 mg daily for 1 year
  Arms: Moderate-dose statin therapy

SUMMARY:
During coronary artery bypass graft surgery (CABG), saphenous vein from the leg is used to bypass the atherosclerotic blockages in the arteries of the heart. Unfortunately, vein bypasses themselves develop blockages over time, a process termed saphenous vein graft disease. By lowering cholesterol levels in the blood, statin medications are used after surgery to prevent the development of atherosclerotic blockages in the vein bypasses. Recently, higher doses of statin medications have been introduced, with some studies showing that they are more effective than traditional doses when used in heart attack patients. Furthermore, laboratory tests have shown that higher doses of statin medications can slow the development of atherosclerosis. Despite these benefits, very little is known regarding the use of high-dose statin therapy after bypass surgery in humans.

The goal of this study will be to see if high-dose statin therapy will prevent the development of vein graft occlusion during the first year after bypass surgery. Patients will be randomized to receive either high-dose statin therapy or conventional moderate-dose statin therapy starting within 4 days of surgery and continuing for the duration of one year after the operation. The statin medication will be given in capsule form. During the course of this study, neither the patient nor the health care team will know which treatment each patient is receiving. One year after bypass surgery, a computed tomography (CT) coronary angiogram will be performed to evaluate the patency of the vein bypasses.

DETAILED DESCRIPTION:
The current clinical guidelines recommend treatment to achieve LDL levels <100 mg/dL after surgical coronary revascularization. However, recent studies have illustrated that even more intensive lipid reduction with high-dose statins can further improve cardiovascular outcomes. Targeting LDL levels to 70 mg/dL after CABG with intensive statin therapy may prevent the process of postoperative saphenous vein graft disease and lead to improved graft patency. Therefore, in the ACTIVE Trial, we will conduct a randomized controlled trial comparing high-dose (80 mg atorvastatin) to moderate-dose (10 mg atorvastatin)statin therapy in patients undergoing CABG with saphenous vein grafts. The effect of aggressive cholesterol therapy on the process of vein graft disease will be examined with computed tomography (CT) coronary angiography one year after CABG. This study will address the subject of postoperative high-dose statin therapy and help determine the optimal lipid-lowering strategy following CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first-time CABG with at least 1 saphenous vein graft

Exclusion Criteria:

* Redo-CABG
* Statin allergy
* Severe renal dysfunction
* Severe liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2012-03; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kulik, MD MPH, Principal Investigator — Lynn Heart and Vascular Institute, Boca Raton Regional Hospital; Marc Ruel, MD MPH, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Lynn Heart and Vascular Institute, Boca Raton Regional Hospital, Boca Raton, Florida, United States
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kulik A, Voisine P, Mathieu P, Masters RG, Mesana TG, Le May MR, Ruel M. Statin therapy and saphenous vein graft disease after coronary bypass surgery: analysis from the CASCADE randomized trial. Ann Thorac Surg. 2011 Oct;92(4):1284-90; discussion 1290-1. doi: 10.1016/j.athoracsur.2011.04.107. PMID 21958773
- [Background] Kulik A, Ruel M. Lipid-lowering therapy and coronary artery bypass graft surgery: what are the benefits? Curr Opin Cardiol. 2011 Nov;26(6):508-17. doi: 10.1097/HCO.0b013e32834b9fb1. PMID 21934497
- [Background] Kulik A, Ruel M. Statins and coronary artery bypass graft surgery: preoperative and postoperative efficacy and safety. Expert Opin Drug Saf. 2009 Sep;8(5):559-71. doi: 10.1517/14740330903188413. PMID 19673591
- [Derived] Kulik A, Abreu AM, Boronat V, Ruel M. Intensive versus moderate atorvastatin therapy and one-year graft patency after CABG: Rationale and design of the ACTIVE (Aggressive Cholesterol Therapy to Inhibit Vein Graft Events) randomized controlled trial (NCT01528709). Contemp Clin Trials. 2017 Aug;59:98-104. doi: 10.1016/j.cct.2017.06.006. Epub 2017 Jun 10. PMID 28611006

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-dose Statin Therapy | Moderate-dose Statin Therapy
Started | 86 | 87
Completed | 73 | 72
Not Completed | 13 | 15
Not completed — Death | 2 | 0
Not completed — Withdrawal by Subject | 10 | 15
Not completed — allergy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-dose Statin Therapy | Moderate-dose Statin Therapy | Total
Number analyzed (Participants) | 86 | 87 | 173
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.4) | 70.5 (10.4) | 68.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 73 | 68 | 141
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diabetes [Count of Participants; unit: Participants] | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Saphenous Vein Graft Occlusion (Percentage of Vein Grafts Occluded) Based on CT Coronary Angiography at 1 Year
Description: Vein graft patency will be assessed in a blinded fashion by CT coronary angiography 1 year after CABG
Time Frame: 1 year after CABG
Measure: Count of Units; unit: Vein grafts
Units Other Than Participants: Vein grafts
Arm/Group | High-dose Statin Therapy | Moderate-dose Statin Therapy
Number analyzed (Participants) | 73 | 72
Number analyzed (Vein grafts) | 123 | 124
Vein grafts | 14 | 16

2. Secondary Outcome: Vein Graft Stenosis 1 Year After CABG Based on CT Coronary Angiography
Description: Vein graft stenosis 1 year after CABG based on CT coronary angiography
Time Frame: Within 1 year after CABG
Measure: Count of Units; unit: Vein grafts
Units Other Than Participants: Vein grafts
Arm/Group | High-dose Statin Therapy | Moderate-dose Statin Therapy
Number analyzed (Participants) | 73 | 72
Number analyzed (Vein grafts) | 123 | 124
Vein grafts | 4 | 7

ADVERSE EVENTS:
Arm/Group | High-dose Statin Therapy | Moderate-dose Statin Therapy
All-Cause Mortality (participants affected / at risk) | 2/86 | 0/87
Serious Adverse Events (participants affected / at risk) | 5/86 | 7/87
Other Adverse Events (participants affected / at risk) | 0/86 | 0/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High-dose Statin Therapy (N=86) | Moderate-dose Statin Therapy (N=87)
Uncontrolled lipid levels (Metabolism and nutrition disorders) | 2 | 6
Elevated CK levels (Musculoskeletal and connective tissue disorders) | 0 | 1
Elevated liver enzymes (Hepatobiliary disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No